CLINICAL TRIAL: NCT00303160
Title: Effect of Helicobacter Pylori on the Availability of Vitamin E and C
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: CCERN: canadian cancer etiology research network (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15344
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2007-08-14 (Estimated); Status verified 2007-08

CONDITIONS: Heliobacter Pylori Infection
Keywords: heliobacter pylori infection; reactive oxygen species; antioxidants
MeSH Terms: interventions — Ascorbic Acid

INTERVENTIONS:
Drug: vitamin C & E supplements

SUMMARY:
This study argues that H.pylori infection, by increasing the production of reactive oxygen species, increases the utilization of dietary antioxidants(Vit E and Vit C) that serve in quenching the free radicals, thus decreasing their serum levels and confounding their protective effect against gastric cancer.

DETAILED DESCRIPTION:
It has been postulated that dietary antioxidants may reduce cancer risk by modulating red-ox status, by preventing biological oxidation, and by inhibiting the formation of carcinogen. However, supplementation studies and prospective studies have yielded contradictory results. In the case of gastric cancer, H.pylori infection, which is known to be associated with a higher risk of the disease, results in an increased production of ROS & RNS. As a result serum levels of these free radicals increase, exerting a higher demand for dietary antioxidants to neutralize them.

The fact that the relation between serum levels of antioxidants and gastric cancer is more consistent than that of dietary intake levels and the disease suggests the possibility of the presence of an intrinsic factor that is altering the true relation between dietary antioxidants and the cancer. This intrinsic factor, this study argues, is the infection with H.pylori.

H.pylori infection, by increasing the production of reactive oxygen species, increases the utilization of dietary antioxidants that serve in quenching the free radicals, thus decreasing their serum levels and confounding their protective effect against gastric cancer. The purpose of this pilot study is to investigate the possibility that H.pylori infection alters the bioavailability of the dietary antioxidants: vitamin C, and vitamin E. This project will be done in preparation for an etiologic study of dietary antioxidants and gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult , age 18-45

Exclusion Criteria:

1. Smoking
2. Body mass index below 18 or above 25.
3. Previous treatment for H.pylori infection
4. Partial or total gastrectomy
5. History of gastritis
6. Currently taking antioxidants supplementation
7. Training in an athletic team.
8. Drinking more than 3 servings of alcohol/day

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2006-03; Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
plasma vitamin C levels
plasma vitamin E levels

SECONDARY OUTCOMES:
TBARS levels

CONTACTS AND LOCATIONS:
Overall Officials: Farah Naja, MSc., Principal Investigator — Canada: Cancer Care Ontario
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada